#### The GlaxoSmithKline group of companies

| Division | Worldwide Development |
|------------------|-----------------------------------|
| Information Type | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for 206243, A Prospective,<br>Longitudinal Study to Investigate the Effect of Thermal<br>Injury on Intestinal Permeability and Systemic Inflammation<br>(HESTIA). |
|---|---|---|
| Compound Number | : | No Compound |
| Effective Date | : | 27-NOV-2018 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206243.
- This RAP is intended to describe the planned safety and Biomarker analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.

## Author(s)

| Author | |
|------------|-------------------------------------|
| Lead | PPD |
| | Statistics Leader (Biostatistics) |
| Co-Authors | PPD |
| | Senior Statistician (Biostatistics) |

# RAP Team Review Confirmations (Method: E-mail)

| Reviewer | Date |
|--------------------------------------|-------------|
| Associate Programmer (Biostatistics) | 20-NOV-2018 |
| Director (Clinical Development) | 17-NOV-2018 |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date |
|---------------------------------------------------|-------------|
| Senior Statistics Director (Biostatistics) | 27-NOV-2018 |
| Biostatistics Programming Manager (Biostatistics) | 27-NOV-2018 |

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | SUMN | MARY OF | KEY PROTOCOL INFORMATION | 5 |
| •• | 1.1. | | s to the Protocol Defined Statistical Analysis Plan | |
| | 1.2. | | bjective(s) and Endpoint(s) | |
| | | 1.2.1. | Protocol Defined Objectives and Endpoints | |
| | | 1.2.2. | Final Reporting Objectives & Endpoints Following Study | |
| | | | Termination | |
| | 1.3. | • | esign | |
| | 1.4. | Statistica | al Hypotheses / Statistical Analyses | 8 |
| 2. | | | LYSES | |
| | 2.1. | | Analyses | |
| | 2.2. | Final An | alyses | 9 |
| 3. | ANAL | | PULATIONS | |
| | 3.1. | Protocol | Deviations | 9 |
| 4. | CONS | SIDERATION | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | | S | |
| | 4.1. | | Considerations | |
| | 4.2. | | Definitions | |
| | | 4.2.1. | Derivations and Handling of Missing Baseline Data | 12 |
| 5. | STUD | | ATION ANALYSES | |
| | 5.1. | Overviev | w of Planned Study Population Analyses | 13 |
| 6. | EFFIC | ACY ANA | ALYSES | 13 |
| | 6.1. | | Analyses | |
| | | 6.1.1. | Endpoint / Variables | |
| | | 6.1.2. | Summary Measure | |
| | | 6.1.3. | Population of Interest | |
| | | 6.1.4. | Statistical Analyses / Methods | |
| | 6.2. | • | ory Analyses | |
| | | 6.2.1. | Endpoint / Variables | |
| | | 6.2.2. | Summary Measure | 13 |
| | | 6.2.3. | Population of Interest | 14 |
| | | | 6.2.3.1. Statistical Analyses / Methods | 14 |
| | | | 6.2.3.2. Statistical Methodology Specification | 14 |
| 7. | SAFF | TY ANAL` | YSES | 15 |
| | 7.1. | | Events Analyses | |
| | 7.2. | | Laboratory Analyses | |
| | 7.3. | | afety Analyses | |
| _ | | | | |
| 8. | | | NALYSES | |
| | 8.1. | | ory Biomarker Analyses | |
| | | 8.1.1. | Endpoint / Variables | |
| | | 8.1.2. | Summary Measure | |
| | | 8.1.3. | Population of Interest | |
| | | | 8.1.3.1. Statistical Analyses / Methods | 16 |

#### CONFIDENTIAL

| | | | 8.1.3.2. | Statistical Methodology Specification | 17 |
|---|---|---|---|---|---|
| 9. | REFE | RENCES. | | | 18 |
| 10. | | | | | |
| | 10.1. | Appendi | | ule of Activities | |
| | | 10.1.1. | | Defined Schedule of Events | |
| | 10.2. | | | sment Windows | 23 |
| | 10.3. | | | Phases and Treatment Emergent Adverse | |
| | | 10.3.1. | | ases | |
| | | | | Study Phases for Concomitant Medication | |
| | 10.4. | | | isplay Standards & Handling Conventions | |
| | | 10.4.1. | | Process | |
| | | 10.4.2. | - 1 | Standards | |
| | 10.5. | | | d and Transformed Data | |
| | | 10.5.1. | | | |
| | | 10.5.2. | | | |
| | | 10.5.3. | | | |
| | 10.6. | | | ing Standards for Missing Data | |
| | | 10.6.1. | | e Withdrawals | |
| | | 10.6.2. | | of Missing Data | |
| | | | | Handling of Missing and Partial Dates | |
| | 10.7. | | | viations & Trade Marks | |
| | | 10.7.1. | | ions | |
| | | 10.7.2. | | ks | |
| | 10.8. | | | Data Displays | |
| | | 10.8.1. | | lay Numbering | |
| | | 10.8.2. | | imple Shell Referencing | |
| | | 10.8.3. | | les | |
| | | 10.8.4. | | oulation Tables | |
| | | 10.8.5. | , | ables | |
| | | 10.8.6. | | igures | |
| | | 10.8.7. | • | bles | |
| | | 10.8.8. | | r Tables | |
| | | 10.8.9. | | r Figures | |
| | | | | gs | |
| | | | | Listings | |
| | 10.9. | Appendi | x 9: Examp | ole Mock Shells for Data Displays | 43 |

## 1. SUMMARY OF KEY PROTOCOL INFORMATION

# 1.1. Changes to the Protocol Defined Statistical Analysis Plan

This study was terminated prior to the full sample size being achieved. As a result the initially planned sample size of 25 for the thermally injured subjects is greatly reduced to 3. Changes from the originally planned statistical analysis specified in the protocol (Dated:26SEP2017) are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Pro | Protocol | | Reporting & Analysis Plan | | |
|---|---|---|---|---|---|
| Sta | tistical Analysis Plan | | Statistical Analysis Plan | | Rationale for Changes |
| • | Co -Primary Objective 1: To determine the impact of thermal injury on the magnitude of small intestinal permeability change as soon as possible following injury compared to healthy participants. | • | Summary statistics for Lactulose/Mannitol (L/M) ratio at entry will be provided. No formal stats analysis for comparing the groups. | • | No stats analysis due to limited sample size. |
| • | Exploratory objective 1: Comparison of Fractional excretion of sucralose of TI participants with Healthy participants at baseline | • | Only summary will be provided. No formal stats analysis for comparing the groups. | • | No stats analysis due to limited sample size. |
| • | <ul> <li>Exploratory objective 3:</li> <li>Number of ventilator-free days, vasopressor-free days, hemofiltration-free days, episodes of confirmed infection and sepsis, surgical interventions</li> <li>Total length of hospital stay</li> <li>Calculate critical care and thermal injury severity scores</li> </ul> | • | None of the endpoints will be analysed for final reporting. | | <ul> <li>Due to limited sample size, these endpoints will not be analysed.</li> <li>Where relevant, these will be described using data from the SIFTI2 CRF in CSR.</li> </ul> |
| • | Exploratory objective 4: Change in urine protein: creatinine and urine albumin: creatinine ratios | • | This endpoint will not be analysed. | • | The reason for collecting these data was to inform a pharmacokinetic model. As development of the molecule has been terminated, this model is no longer required, moreover data collected are so limited that analysis is not possible. |
| • | Exploratory objective 5:<br>Changes in microbiome of acute and<br>convalescent stool samples | • | This endpoint is not considered for final analysis. | • | Only one stool sample has been collected from a TI patient thus no meaningful comparison is possible. |
| • | Exploratory objective 7:<br>Time to wound recovery | • | This endpoint will not be analysis but will be listed. | • | Sufficient data not available to perform the analysis. |
| • | Exploratory objective 8: • Determine fluid input/output balance | • | These endpoints are not considered for final | • | Sufficient data not available to perform the analysis. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| over time • Changes in serum albumin and plasma creatinine | analysis. | |
| <ul> <li>Exploratory objective 9:</li> <li>Changes in intestinal microbiome</li> <li>Bacterial markers of translocation</li> </ul> | <ul> <li>No microbiome data<br/>analysis</li> <li>Bacterial markers of<br/>translocation will be<br/>summarised.</li> </ul> | Insufficient stool samples<br>have been collected for<br>correlative analyses in TI<br>participants. |

# 1.2. Study Objective(s) and Endpoint(s)

# 1.2.1. Protocol Defined Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To determine the impact of thermal injury on the<br>magnitude of small intestinal permeability change as<br>soon as possible following injury compared to health<br>participants | |
| To characterise the effect of thermal injury on small intestinal permeability over time and establish the clinical and demographic factors which can influence it | |
| Exploratory Objectives | Exploratory Endpoints |
| To determine the impact of thermal injury on colonic<br>permeability as soon as possible following injury<br>compared to healthy participants | Fractional excretion of sucralose at entry |
| To characterise the effect of thermal injury on coloni permeability over time | Changes in the fractional excretion of sucralose over time |
| To assess the relationship between severity of a participant's condition following thermal injury and | Number of ventilator-free days |
| changes in intestinal permeability | Number of vasopressor-free days |
| | Number of hemofiltration-free days |
| | <ul> <li>Number of episodes of confirmed infection<br/>and sepsis</li> </ul> |
| | <ul> <li>Number of surgical interventions</li> </ul> |
| | Total length of hospital stay |
| | <ul> <li>Calculate critical care and thermal injury severity scores</li> </ul> |
| To assess plasma and urine biomarkers of intestinal<br>permeability, bacterial translocation and renal tubular | |
| dysfunction following thermal injury | Change in urine protein: creatinine and urine albumin: creatinine ratios |
| To assess the impact of thermal injury and intestinal permeability on the intestinal microbiome compared | |

| Objectives | Endpoints |
|---|---|
| to healthy participants | convalescent stool samples |
| To assess the impact of pre-existing co-morbid conditions on intestinal permeability and clinical outcome following thermal injury | Medical history and drug history at the time of admission |
| To assess wound healing | Time to wound recovery (e.g. 95%) |
| To characterise parameters that may influence drug PK/PD | Determine fluid input/output balance over time |
| | Changes in serum albumin and plasma creatinine |
| To characterise intestinal microbiota, and correlate its composition with both intestinal permeability and bacterial detection in blood | <ul> <li>Changes in intestinal microbiome</li> <li>Bacterial markers of translocation</li> </ul> |

# 1.2.2. Final Reporting Objectives & Endpoints Following Study Termination

| | jectives | Endpoints |
|---|---|---|
| Pri | mary Objectives | Primary Endpoints |
| • | To determine the impact of thermal injury on the magnitude of small intestinal permeability change as soon as possible following injury compared to healthy participants | Lactulose/Mannitol (L/M) ratio at entry |
| • | To characterise the effect of thermal injury on small intestinal permeability over time and establish the clinical and demographic factors which can influence it | Changes in L/M ratio over time |
| Ex | ploratory Objectives | Exploratory Endpoints |
| • | To determine the impact of thermal injury on colonic permeability as soon as possible following injury compared to healthy participants | Fractional excretion of sucralose at entry |
| • | To characterise the effect of thermal injury on colonic permeability over time | Changes in the fractional excretion of sucralose over time |
| • | To assess plasma and urine biomarkers of intestinal permeability and bacterial translocation | Change in markers of intestinal mucosal damage samples from blood |
| | | Change in bacterial markers of translocation |
| • | To assess the impact of pre-existing co-morbid conditions on intestinal permeability and clinical outcome following thermal injury | Medical history and drug history at the time of admission |

## 1.3. Study Design



Note: The above design was prior to study termination. The study was terminated before any subjects had reached day 28. Hence, later visits are not included in the analysis.

# 1.4. Statistical Hypotheses / Statistical Analyses

- No formal hypothesis testing is planned.
- The key factors of interest in this study were to understand (i) the nature of any differences at entry in intestinal permeability between healthy participants and thermal injury participants (ii) to understand the trajectory of changes in intestinal permeability over time.

## 2. PLANNED ANALYSES

### 2.1. Interim Analyses

No formal interim analysis will be performed.

## 2.2. Final Analyses

The analyses will be performed after completion of the following sequential steps:

- 1. All subjects have completed Day 28 assessments or have withdrawn from the study.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All protocol deviations have been confirmed.
- 4. Analysis population exclusions have been confirmed.
- 5. Database freeze has been declared by Data Management.

#### 3. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul><li>Study Population</li><li>All Listings</li></ul> |
| Safety | Comprise of all participants who receive at least<br>one dose of STM and have at least one post-dose<br>safety assessment. | Safety |
| Evaluable | Comprises of all participants in the safety population excluding any healthy volunteers that received any concomitant medication or food and drink containing STM (lactulose, mannitol and sucralose), as identified by review of the protocol deviations. | <ul><li>Efficacy</li><li>Biomarker</li><li>Study Population</li></ul> |

#### NOTES:

 Please refer to Appendix 8: List of Data Displays which details the population to be used for each display being generated.

#### 3.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

Prospective approval of protocol deviations to recruitment and enrolment criteria, also known as protocol waivers or exemptions, is not permitted.

# 4. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 2 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 2 Overview of Appendices

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Assessment Windows |
| 10.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Reporting Standards for Missing Data |
| 10.7 | Appendix 7: Abbreviations & Trade Marks |
| 10.8 | Appendix 8: List of Data Displays |
| 10.9 | Appendix 9: Example Mock Shells for Data Displays |

#### 4.1. General Considerations

• This is a longitudinal, prospective study of healthy participants and participants who have sustained thermal injury.

#### Unless otherwise stated, the following rules will apply:

- Summaries and displays will be presented by study group and visit (without the group information in visit).
- The following statistics will be used to summarise the data, unless otherwise specified:
  - o Continuous Variables: number of observations (n), mean, standard deviation (SD), standard error (SE), median, minimum and maximum.
  - Categorical Variables: number of observations (n), frequency counts and percentages.
- Summaries by Visit: Only scheduled visits will be presented, unless otherwise stated. Unscheduled visits will be listed but will not contribute towards any summary statistics/analyses, unless otherwise stated.
- Summaries by study group: Study group (Healthy Participants and TI Participants) will be used instead of treatment group in all the tables and listing.
- No imputation will be done for missing values across visits, individual missing scores will be considered missing.

#### 4.2. Baseline Definitions

For efficacy and biomarker endpoints, the baseline value will be Day 1 for both the groups. In case of missing Day 1 assessment, baseline would be set to missing.

| Parameter | <u> </u> | Study Assessments Considered as<br>Baseline | |
|---|---|---|---|
| | Screening [1] | Day 1 (Baseline) | |
| Efficacy Assessments | | | |
| L/M Ratio | | X | Day 1 (Baseline) |
| Fractional excretion of sucralose | | X | Day 1 (Baseline) |
| Biomarkers Assessments | | | |
| Markers of intestinal mucosal damage | | X | Day 1 (Baseline) |
| Bacterial markers of translocation | | X | Day 1 (Baseline) |
| Safety Assessments | | | |
| Vital Signs | Χ | | Screening |
| Laboratory Assessments | | | |
| Haematology | Χ | | Screening |
| Clinical Chemistry | Х | | Screening |
| Routine Urinalysis | Χ | | Screening |
| [1] Screening = 1-2 Wks Prior to Day 1 (Heal | [1] Screening = 1-2 Wks Prior to Day 1 (Healthy Participants). | | |

### 4.2.1. Derivations and Handling of Missing Baseline Data

For untransformed data, change from baseline at each time point is expressed as a difference (value at time point – value at baseline).

| Definition | Reporting Details |
|---|---|
| Change from Baseline [1] | = Post-Baseline Visit Value – Baseline Value |
| % Change from Baseline [1] | = 100 x [(Post-Baseline Visit Value – Baseline Value) / Baseline Value] |
| [1] If the baseline value is missing the change from baseline derivations will also be missing | |

#### 5. STUDY POPULATION ANALYSES

## 5.1. Overview of Planned Study Population Analyses

• The Study Population analyses will be based on the Screened, Evaluable or Safety population, as appropriate unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 8: List of Data Displays.

#### 6. EFFICACY ANALYSES

## 6.1. Primary Analyses

#### 6.1.1. Endpoint / Variables

• Lactulose/mannitol ratio

### 6.1.2. Summary Measure

The administration of the STM is for the purpose of intestinal permeability measurement and is not therapeutic, therefore no efficacy will be assessed.

Absolute, change and % change in lactulose/mannitol ratio values will be used for analysis.

#### 6.1.3. Population of Interest

The primary analyses will be based on the evaluable population, unless otherwise specified.

#### 6.1.4. Statistical Analyses / Methods

Endpoints defined in Section 6.1.1 will be summarised by study group, timepoint and visit. Data will summarise mean, standard deviation, standard error, minimum, median, maximum and N.

No formal statistical analysis will be performed.

#### 6.2. Exploratory Analyses

#### 6.2.1. Endpoint / Variables

• Fractional excretion of sucralose

#### 6.2.2. Summary Measure

Absolute, Change and %Change in the fractional excretion of sucralose over

time.

## 6.2.3. Population of Interest

The exploratory efficacy analyses will be based on the evaluable population, unless otherwise specified.

#### 6.2.3.1. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints defined in Section 6.2.1 will be summarised using descriptive statistics and listed.

#### 6.2.3.2. Statistical Methodology Specification

There will be no planned statistical analysis.

#### 7. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 8: List of Data Displays.

NOTE: As detailed in Section 9.2.1 of the protocol, only AEs deemed to be related to procedures or requirements unique to the HESTIA study will be recorded/reported for thermally injured participants. All other AEs will be recorded/reported through the SIFTI-2 study.

Also, as given in Section 12.4 (Events NOT Meeting the AE Definition) in protocol, any clinically significant abnormal laboratory findings or other abnormal safety assessments which are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition will be considered as disease related event. Table 3 in protocol provides a list of commonly occurring AEs in participants with severe thermal injury which may meet this definition and will be entered as disease related events.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests and Urinalysis will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 8: List of Data Displays.

Table 3 Protocol-Required Safety Laboratory Assessments for Healthy Participants:

| Laboratory<br>Assessments | Parameters | | | | |
|---|---|---|---|---|---|
| | Platelet Count | | WBC count with Differential: | | |
| Hematology | RBC Count | | Neutrophils<br>Lymphocytes | | |
| riomatology | Hemoglobin | | Monocytes<br>Eosinophils | | |
| | Hematocrit | | | Basophils | |
| | Urea | Potassium | | | Total bilirubin |
| Clinical Chemistry | Creatinine | Sodium | Alanine Amin<br>(ALT) | otransferase | Total Protein |
| , | Glucose non-<br>fasting | Calcium | phatase | | |
| Routine Urinalysis | pH, glucose, protein, blood, ketones by dipstick Microscopic examination (if blood or protein is abnormal) | | | | |

### 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 8: List of Data Displays.

#### 8. BIOMARKER ANALYSES

### 8.1. Exploratory Biomarker Analyses

### 8.1.1. Endpoint / Variables

As this is an exploratory study, a number of data presentations will be produced for a set of biomarkers to understand how they change over time. In order to simplify the investigation, the biomarkers will be grouped into biomarkers of intestinal damage and bactorial markers of translocation. All endpoints will be summarised by mean, standard deviation, standard error, median, minimum, maximum and number of subjects, by study group. These groupings of biomarkers are provided in Table 4.

Table 4 List of biomarkers considered for final analysis

| Biomarker Grouping | Parameters |
|---|---|
| Markers of intestinal mucosal damage | iFABP, citrulline, Zonulin-1, Occludin |
| Bacterial markers of translocation | sCD14, Microbial Metabolites: (Glycodeoxycholic acid, Taurodeoxycholic acid, Taurodeoxycholic acid, Taurolithocholic acid, Oxocholic acid, Ursodeoxycholic acid) |

#### 8.1.2. Summary Measure

- Change in markers of intestinal mucosal damage samples from blood.
- Changes in Bacterial markers of translocation.

#### 8.1.3. Population of Interest

The exploratory efficacy analyses will be based on the evaluable population, unless otherwise specified.

#### 8.1.3.1. Statistical Analyses / Methods

Unless otherwise specified, endpoints defined in Section 8.1.1 will be summarised using descriptive statistics and listed.

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

# 8.1.3.2. Statistical Methodology Specification

There will be no planned statistical analysis.

## 9. REFERENCES

GlaxoSmithKline Document Number 2016N289648\_02, Study ID 206243/02, A Prospective, Longitudinal Study to Investigate the Effect of Thermal Injury on Intestinal Permeability and Systemic Inflammation (HESTIA). Effective Date: 26-SEP-2017.

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

## 10.1.1. Protocol Defined Schedule of Events

## **Healthy Participants (Group 1)**

| Procedure | Screening | Treatment P | eriod [Out pat<br>1 day) | Notes | |
|---|---|---|---|---|---|
| | | D1 | D8 | D15 | |
| Review of inclusion/ exclusion criteria and informed consent | X | | | | |
| Demography | X | | | | |
| Medical history (includes substance and alcohol usage at screening) and Medication history | X | | | | |
| Substance testing (urine) | X | | | | Substances: [Recreational Drugs and Alcohol] |
| HIV, Hepatitis B and C screening | X | | | | If test otherwise performed within 3 months prior to study entry, testing is not required |
| Laboratory assessments | X | | | | |
| Pregnancy test (WOCBP only) (urine) | X | (X) | | | Only performed again on Day 1 if patient at risk of pregnancy at or since screening |
| Blood sampling for biomarkers | | X | | | 20ml of blood will be sampled in a single draw on one day, preferably Day 1 |
| Stool sample collection | | X | | | Participants will be given a collection container at screening to bring with them on Day 1. |
| Brief physical examination including measurements of height and weight Vital Signs (systolic and diastolic blood | X | X | X | X | BMI calculated from height and weight at screening only Examinations should be conducted the day after intestinal permeability measurement. |
| pressure and heart rate) Medical review (assessment of health status) | | X | X | X | Monitor for signs and symptoms of gastro-intestinal infections and other emergent issues |

| Procedure | Screening | Treatment Po | eriod [Out pat<br>1 day) | Notes | |
|---|---|---|---|---|---|
| | | D1 | D8 | D15 | |
| STM Training | X | | | | Refresher training may be provided as needed |
| Intestinal permeability measurement: | | | | | Please refer to SRM for full information |
| STM administration followed by a 24- | | X | X | X | Intestinal permeability measurement to be performed |
| hour urine collection | | | | | at home the day before the study visit. |
| AE/SAE and Concomitant medication | (V) | , | | 、 | Day 1 will include concomitant medication review |
| reviews | (X) | <b>——</b> | | → | only |

**Thermal Injury Participants (Group 2)** 

| 0 | | Treatment Period [ICU Days] (+/4 hours) | | | | | | | 6 mon | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | D1<br>(≤ 24 hr of<br>admission) | D2 | D3 | D4 | D5 | D6 | D7 | D8 | D9 | D<br>10 | D<br>11 | D<br>12 | D<br>13 | D<br>14 | D28 (± 3 days) | (± 14<br>days) | Notes |
| Review of inclusion/ exclusion criteria and informed consent | X | | | | | | | | | | | | | | | | Participants will be co-<br>consented to the SIFTI-2<br>study |
| Medical history<br>(includes substance<br>and alcohol usage)<br>and Medication<br>history | X | | | | | | | | | | | | | | | | |
| Substance testing (urine) | X | | | | | | | | | | | | | | | | Substances: [Recreational Drugs, Alcohol] |
| Pregnancy test<br>(WOCBP only)<br>(urine) | X | | | | | | | | | | | | | | | X | To be repeated at 6 months prior to final STM administration |
| HIV, Hepatitis B and C screening | X | | | | | | | | | | | | | | | | If test otherwise performed within 3 months prior to study entry, testing is not required |
| Initial assessment of Burns | X | | | | | | | | | | | | | | | | Calculation of %TBSA Location of thermal injury and depth |
| Fluid balance (total input/output) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X* | | Daily (over 24 hr) *only if participant still admitted |
| Intestinal permeability measurement: STM administration followed by a 24- hour urine collection | X | | X | | X | | X | | X | | X | | X | | Х | X | Measurements every 48 hours from first measure. Preference: D1, 3, 5, 7, 9, 11, 13. Otherwise: D2, 4, 6, 8, 10, 12, 14. Please refer to SRM for full method. |

| Brief Physical<br>Examination | | | | | | | | X | X | Following final intestinal permeability measurement. Can be omitted if patient is still admitted to hospital. |
|---|---|---|---|---|---|---|---|---|---|---|
| Stool sample collection | | (A | $\leftarrow = \Rightarrow \qquad \qquad X \qquad X$ (A sample of the first stool produced following admission) | | | X | Time to first stool collection;<br>preferably on Day 1. Then on<br>Days 14 and 28 and 6<br>months | | | |
| Wound Healing<br>Assessments | | | | | | | X | X | X | This is to assess time to 95% wound healing |
| AE/SAE and<br>Concomitant<br>medication reviews | X | ←=============== | | X | AE/SAE monitoring will<br>begin after the first<br>administration of STM | | | | | |

Planned time points for all safety assessments are provided in the SoA and summarised here.

| | When conducted | |
|---|---|---|
| Safety Assessment | Healthy Participants | Thermally injured participants |
| Laboratory tests | Screening. Only repeated if clinically indicated in the opinion of the investigator. | Only if clinically indicated. |
| Brief Physical Examination including Vital Signs Recording | Screening, Day 1, Day 8, Day 15 | As a part of routine clinical care whilst admitted (not protocol specified). Following day 28 and 6-month intestinal permeability measurements (if patient not still admitted) |
| <b>Detection of AEs</b> | Day 1, Day 8, Day 15 | Throughout the study |
| Assessment of health status | Screening, Day 1, Day 8, Day 15 | Not required |

# 10.2. Appendix 2: Assessment Windows

No visit slotting will be done.

# 10.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 10.3.1. Study Phases

### 10.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

### NOTES:

• Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

#### 10.4.1. Reporting Process

| Software | |
|---|---|
| The currently support | The currently supported versions of SAS software 9.4 or higher will be used. |
| Reporting Area | |
| HARP Server | : Uk1salx00175\arprod\nocompound\mid206243 |
| HARP Compound | : No Compound |
| QC Spreadsheet : Uk1salx00175\arwork\nocompound\mid206243\Documents | |
| Analysis Datasets | Analysis Datasets |
| Analysis datasets will be created according to IDSL standards. | |
| Generation of RTF Files | |
| RTF files will be generated for SAC. | |

### 10.4.2. Reporting Standards

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### CONFIDENTIAL

| Unscheduled Visits | Unscheduled Visits |
|---|---|
| Unscheduled visits | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled vi | All unscheduled visits will be included in listings. |
| Descriptive Summary | Descriptive Summary Statistics |
| Continuous Data | Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.

#### **Study Day**

- Calculated as the number of days from First STM Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First STM Dose Date → Study Day = Ref Date First STM Dose Date</li>
  - Ref Data ≥ First STM Dose Date → Study Day = Ref Date (First STM Dose Date) + 1

#### Age

Age = Screening date – Date of Birth
 Date of birth will be imputed based on the assumption that all subjects were born on the 30th June (30 Jun YYYY).

#### Baux score

Baux score: Age + % Total Body Surface Area (TBSA) burned

#### 10.5.2. **Efficacy**

#### Fractional Excretion of Lactulose/Mannitol/Sucralose

Data is provided to S&P in the form of quantity of material in micrograms/litre, based on a sample of urine.

Fractional excretion (FE) of lactulose or mannitol or sucralose = (urine concentration (micrograms/litre) × total urine volume excreted in litre) / probe input (micrograms).

#### Where,

- Urine concentration is provided in the BIOMARKER dataset,
- Urine volumes excreted are provided in the BIOLINK dataset,
- Probe input refers to the total STM taken (as per Table 7.1 of the protocol-5g Lactulose, 2g Mannitol and 2g Sucralose)

Urine concentration in the BIOMARKER dataset will be provided at two timepoints per visit (0-5hr) and (0-24hr)

FE will be calculated for timepoints 0-5 and 0-24 hours for Lactulose, Mannitol and Sucralose.

For calculations of the 0-24 FE's, total urine volume will be based on the following:

Total urine=urine excreted 0-5 hrs + urine excreted 5-24 hours.

Note: If urine excreted 0-5 hrs is missing then total urine should be considered missing.

Note: 1g=1000000 micrograms

#### L/M ratio

L/M ratio = FE lactulose / FE mannitol

#### **Healthy Participant – Average**

• Average = Mean of all data available at all timepoint for each healthy participant.

### 10.5.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Points = '< x' becomes x 0.01
  - Example 2: 1 Decimal Point = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Points = '< x' becomes x 1

# 10.6. Appendix 6: Reporting Standards for Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as if he/she receives all planned doses of STM and completes the Day 15 in case of healthy participants and 6 months in case of participants with thermal injuries.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |

# 10.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of STM; in this case the STM start date will be used.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of STM; in this case the STM stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> </ul> |
| | Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.7. Appendix 7: Abbreviations & Trade Marks

# 10.7.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ACR | Albumin/creatinine ratio |
| ADaM | Analysis Data Model |
| AE/SAE | Adverse Event/ Serious Adverse Event |
| Anti-HBc | Anti-Hepatitis C |
| ART | Anti-retroviral treatment |
| CDISC | Clinical Data Interchange Standards Consortium |
| CFB | Change from Baseline |
| CFR | Code of Federal Regulations |
| CSR | Clinical Study Report |
| CV | Coefficient of Variation |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| Gl | Gastrointestinal |
| GSK | GlaxoSmithKline |
| НВ | Hepatitis B |
| HBs AG | Hepatitis B Antigen |
| HCV | Hepatitis C |
| HIV | Human Immunodeficiency Virus |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| ICU | Intensive Care Unit |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| ISS | Investigator Sponsored Study |
| L/M | Lactulose/mannitol ratio |
| MODS | Multi-organ dysfunction syndrome |
| NC | Nominated Consultee |
| NIMP | Non-investigational medicinal product |
| PC | Personal Consultee |
| PCR | Polymerase Chain Reaction |
| PDMP | Protocol Deviation Management Plan |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SIFTI-2 | A Multi-centre, Prospective Study to Examine the Relationship between Neutrophil Function and Sepsis in Adults and Children with Severe Thermal Injuries |
| SoA | Schedule of Activities |
| SRM | Study Reference Manual |
| STM | Sugar Test Material |
| TBSA | Total Body Surface Area |
| TI | Thermally Injured |
| TNF | Tumour Necrosis Factor |
| WOCBP | Women of Child Bearing Potential |

# 10.7.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

## 10.8. Appendix 8: List of Data Displays

## 10.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------|------------|
| Study Population | 1.1 to 1.8 | N/A |
| Efficacy | 2.1 to 2.6 | 2.1 to 2.8 |
| Safety | 3.1 to 3.4 | N/A |
| Biomarker | 4.1 to 4.6 | 4.1 to 4.4 |
| Section | List | ings |
| ICH Listings | 1 to | 23 |
| Other Listings | 24 to 27 | |

#### 10.8.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 9: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|---------|
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.8.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.8.4. Study Population Tables

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | | | | |
| 1.1. | Evaluable | ES8 | Subject Status and Reasons for Study Withdrawal | ICH E3, FDAAA, EudraCT. Include study group instead of treatment group. | SAC |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| Protoco | l Deviation | | | | |
| 1.3. | Screened | DV1 | Summary of Important Protocol Deviations | ICH E3. Include study group instead of treatment group. | SAC |
| Populat | ion Analysed | | | | |
| 1.4. | Screened | SP1 | Summary of Study Populations | IDSL. Include study group instead of treatment group. | SAC |
| Demog | raphic and Basel | ine Characteristics | | | |
| 1.5. | Evaluable | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT Add %surface area burnt, Baux score and Body mass index. Include study group instead of treatment group. | SAC |
| 1.6. | Evaluable | DM11 | Summary of Age Ranges | EudraCT Note: Include Age categories: Adult (18 – 64 years), >=65 – 84 years and >=85 years. Include study group instead of treatment group. | SAC |
| 1.7. | Evaluable | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT Include study group instead of treatment group. | SAC |

| Study Po | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell Title Programming Notes | | | | |
| Medical | Medical History | | | | |
| 1.8. | Evaluable | MH4 | Summary of Medical Conditions | ICH E3 Include study group instead of treatment group. Add the medical status (Past/Current). | SAC |

# 10.8.5. Efficacy Tables

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| L/M ratio | L/M ratio | | | | |
| 2.1. | Evaluable | EFF_T1 | Summary of Absolute L/M Ratio Values | Summary by: Study group and Visit Page by: Timepoint | SAC |
| 2.2. | Evaluable | EFF_T1 | Summary of Change in L/M Ratio Values | Note: CFB, Summary by: Study group and Visit, Page by: Timepoint | SAC |
| 2.3. | Evaluable | EFF_T1 | Summary of %Change in L/M Ratio Values | Note: %CFB, Summary by: Study group and Visit, Page by: Timepoint | SAC |
| Fraction | Fractional excretion of sucralose | | | | |
| 2.4. | Evaluable | EFF_T1 | Summary of Fractional Excretion of Sucralose Values | Summary by: Study group and Visit,<br>Page by: Timepoint | SAC |
| 2.5. | Evaluable | EFF_T1 | Summary of Change in Fractional Excretion of Sucralose Values | Note: CFB, Summary by: Study group and Visit, Page by: Timepoint | SAC |
| 2.6. | Evaluable | EFF_T1 | Summary of %Change in Fractional Excretion of Sucralose Values | Note: %CFB, Summary by: Study group and Visit, Page by: Timepoint | SAC |

# 10.8.6. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| L/M ratio | L/M ratio | | | | |
| 2.1. | Evaluable | EFF_F1 | Individual Plot of Absolute L/M Ratio Values Over Time for Healthy Subjects. | Y-axis: Absolute Values Plot by Timepoint | SAC |
| 2.2. | Evaluable | EFF_F2 | Individual Plot of Absolute L/M Ratio Values Over Time for TI Subjects. | Y-axis: Absolute Values Plot by Timepoint Average value of Healthy Subjects will be used as reference line. | SAC |
| 2.3. | Evaluable | EFF_F2 | Individual Plot of %Change L/M Ratio Values Over Time for TI Subjects. | Y-axis: %CFB Values Plot by Timepoint Average value of Healthy subjects will be used as reference. | SAC |
| Fraction | al excretion of s | ucralose | | | |
| 2.4. | Evaluable | EFF_F1 | Individual Plot of Absolute Sucralose Values Over Time for Healthy Subjects. | Y axis: Absolute Values Plot by Timepoint | SAC |
| 2.5. | Evaluable | EFF_F2 | Individual Plot of Absolute Sucralose Values Over Time for TI Subjects. | Y axis: Absolute Values, Plot by Timepoint Average value of Healthy subjects will be used as reference. | SAC |
| 2.6. | Evaluable | EFF_F2 | Individual Plot of %Change Sucralose Values Over Time for TI Subjects. | Y axis: %CFB Values Plot by Timepoint Average value of Healthy subjects will be used as reference. | SAC |

| L/M ratio | L/M ratio and Fractional excretion of sucralose | | | | |
|---|---|---|---|---|---|
| 2.7. | Evaluable | EFF_F3 | Individual Plot of Absolue L/M ratio and Sucralose Values Over Time for TI Subjects. | Y axis: Absolute Values Plot by Timepoint Average values of Healthy subjects will be used as reference. | SAC |
| 2.8. | Evaluable | EFF_F3 | Individual Plot of %Change L/M ratio and Sucralose Values Over Time for TI Subjects. | Y axis: %CFB Values Plot by Timepoint Average values of Healthy subjects will be used as reference. | SAC |

# 10.8.7. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events (AEs) | | | | |
| 3.1. | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 Include study group instead of treatment group. | SAC |
| 3.2. | Safety | AE15 | Summary of Non-Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT Include study group instead of treatment group. | SAC |
| 3.3. | Safety | AE1CP | Summary of Diseases Related Events by Verbatim Term | | SAC |
| Serious and Other Significant Adverse Events | | | | | |
| 3.4. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | SAC |
## 10.8.8. Biomarker Tables

| Pharma | codynamic and | Biomarker: Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Intestin | al Permeability | | | | |
| 4.1 | Evaluable | PD_T1 | Summary of Markers of Intestinal Mucosal Damage | Note: Absolute Values Summary by: Study group and Visit | SAC |
| 4.2 | Evaluable | PD_T1 | Summary of Change in Markers of Intestinal Mucosal Damage | Note: CFB Values<br>Summary by: Study<br>group and Visit | SAC |
| 4.3 | Evaluable | PD_T1 | Summary of % Change in Markers of Intestinal Mucosal Damage | Note: %CFB Values<br>Summary by: Study<br>group and Visit | SAC |
| Bacteria | al Translocation | | | | |
| 4.4 | Evaluable | PD_T1 | Summary of Bacterial Markers of Translocation | Note: Absolute value<br>Summary by: Study<br>group and Visit | SAC |
| 4.5 | Evaluable | PD_T1 | Summary of Change in Bacterial Markers of Translocation | Note: CFB Values<br>Summary by: Study<br>group and Visit | SAC |
| 4.6 | Evaluable | PD_T1 | Summary of % Change in Bacterial Markers of Translocation | Note: %CFB Values<br>Summary by: Study<br>group and Visit | SAC |

# 10.8.9. Biomarker Figures

| Biomar | ker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Biomar | kers | | | | |
| 4.1 | Evaluable | PD_F1 | Individual Plot for Markers of Intestinal Mucosal Damage (Absolute Values) Over Time | Trellis plot – One panel for<br>each biomarker with all TI<br>subjects. Include reference line<br>which is average value of<br>Healthy subjects.<br>Note: Y axis - Absolute Values | SAC |
| 4.2 | Evaluable | PD_F1 | Individual Plot for Markers of Intestinal Mucosal Damage (% Change from baseline Values) Over Time | Trellis plot – One panel for each biomarker with all TI subjects. Include reference line at Zero. Note: Y axis - %CFB Values | SAC |
| 4.3 | Evaluable | PD_F1 | Individual Plot for Bacterial Translocation Associated Biomarkers (Absolute Values) Over Time | Trellis plot – One panel for<br>each biomarker with all TI<br>subjects. Include reference line<br>which is average value of<br>Healthy subjects.<br>Note: Y axis - Absolute Values | SAC |
| 4.4 | Evaluable | PD_F1 | Individual Plot for Bacterial Translocation Associated Biomarkers (% Change from baseline Values) Over Time | Trellis plot – One panel for<br>each biomarker with all TI<br>subjects. Include reference line<br>at Zero Note: Y axis - %CFB<br>Values | SAC |

## **10.8.10. ICH Listings**

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | Screened | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | Screened | SD2 | Listing of Reasons for STM Discontinuation | ICH E3 Mention study group instead of Treatment group. | SAC |
| 4. | Screened | AG1 | Listing of STM administration | | SAC |
| Protoco | ol Deviations | | | | |
| 5. | Screened | DV2 | Listing of Important Protocol Deviations | ICH E3 Mention study group instead of Treatment group. | SAC |
| 6. | Screened | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 Include study group instead of treatment group. | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | tions Analysed | | | | |
| 7. | Screened | SP3 | Listing of Subjects Excluded from Any Population | ICH E3 Mention Evaluable population instead of ITT and per protocol population and study group instead of Treatment group | SAC |
| Demog | raphic and Base | line Characteristics | | | |
| 8. | Screened | DM2 | Listing of Demographic Characteristics | ICH E3 Include study group instead of treatment group. Include Baux score, % surface area burnt and Body mass index. | SAC |
| 9. | Screened | DM9 | Listing of Race | ICH E3 Include study group instead of treatment group. | SAC |
| Conco | mitant Medicatio | ns and Medical Hist | tory | | |
| 10. | Screened | СМЗ | Listing of Concomitant Medications | IDSL Mention study group instead of Treatment group. | SAC |
| 11. | Screened | SU3 | Listing of Substance Use | Include study group instead of treatment group. | SAC |
| 12. | Screened | SP1 | Listing of Subjects Who Had Surgery/Procedure | IDSL Include study group instead of treatment group. | SAC |
| Advers | se Events | | | | |
| 13. | Screened | AE8 | Listing of All Adverse Events | ICH E3 Mention study group instead of Treatment group. | SAC |
| 14. | Screened | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 Include study group instead of treatment group. | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 15. | Screened | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | and Other Sign | ificant Adverse Eve | nts | , | l |
| 16. | Screened | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 Mention study group instead of Treatment group. | SAC |
| 17. | Screened | AE8 | Listing of Disease Related Outcomes/Events. | Only for TI participants. | |
| 18. | Screened | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 Mention study group instead of Treatment group. | SAC |
| 19. | Screened | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 Mention study group instead of Treatment group. | SAC |
| All Lab | oratory | | | | |
| 20. | Screened | LB5 | Listing of All Laboratory Data for all Subjects | ICH E3, Mention study group instead of Treatment group. | SAC |
| 21. | Screened | LB14 | Listing of Laboratory Data with Character Results for all Subjects | ICH E3, Mention study group instead of Treatment group. | SAC |
| 22. | Screened | UR2A | Listing of Urinalysis Data for all Subjects | ICH E3, Include study group instead of treatment group. | SAC |
| Vital Si | gns | | | | |
| 23. | Screened | VS4 | Listing of All Vital Signs Data for all Subjects | IDSL Include study group instead of treatment group. | SAC |

# 10.8.11. Non-ICH Listings

| Non-ICI | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Efficacy | 1 | | | | |
| 24. | Screened | EFF_L1 | Listing of Lactulose, Mannitol, L/M Ratio and Sucralose Data | Note: Numeric Score, CFB & %CFB | SAC |
| Biomar | kers | | | | |
| 25. | Screened | PD_L1 | Listing of Biomarker Data | Note: Include Character result,<br>Numeric score, CFB & %CFB. | SAC |
| Time to | wound recove | ry | | | |
| 26. | Screened | TW_L1 | Listing of Time to Wound Recovery Data for All TI Subjects | | SAC |
| Subject | Characteristic | S | | | |
| 27. | Screened | SC1 | Listing of Subject Characteristics | | SAC |

## 10.9. Appendix 9: Example Mock Shells for Data Displays

Example SP1

Protocol: 206243
Population: Screened

Page 1 of 1

Table 1.5
Summary of Study Populations

| Population | Healthy<br>Subject <b>s</b><br>(N=200) | TI<br>Subjects<br>(N=250) | Total<br>(N=500) |
|---|---|---|---|
| Screened | 200 (100%) | 250 (100%) | 500 (100%) |
| Safety | 195 (98%) | 245 (98%) | 440 (88%) |
| Evaluable | 200 (100%) | 250 (100%) | 460 (92%) |

206243

Page 1 of n

Example EFF\_T1
Protocol: 206243

Population: Evaluable

Timepoint: 0-5 hours/0-24 hours

 $\label{thm:continuous} Table~2.1 \\ Summary~of~Lactulose: Mannitol~(L/M)~ratio~/~Change~in~Lactulose: Mannitol~(L/M)~Ratio~\\ \\$ 

| Study Group | N | Visit | n | Mean | SD | SE | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Healthy<br>Subjects | 200 | Day 1<br>Day 8<br>Day 15<br>Average | 200<br>190<br>186<br>186 | 91.6<br>92.4<br>92.6<br>92.2 | 11.32<br>9.83<br>10.87<br>10.33 | 0.80<br>0.71<br>0.80<br>0.75 | 90.0<br>90.0<br>89.0<br>90.0 | 68<br>70<br>72<br>70 | 140<br>122<br>125<br>140 |
| TI<br>Subjects | 200 | Day 1 Day 3 Day 28 6 months | 200<br>190<br>195<br>186<br>195 | 91.6<br>92.4<br>92.1<br>92.6<br>92.1 | 11.32<br>9.83<br>10.80<br>10.87<br>10.80 | 0.80<br>0.71<br>0.77<br>0.80<br>0.77 | 90.0<br>90.0<br>89.0<br>89.0<br>89.0 | 68<br>70<br>72<br>69<br>72 | 140<br>122<br>120<br>125<br>120 |

Note: Day 1 is considered as baseline for both the study groups.

#### Programming note:

Include all study visits for TI Subjects.

Produce same table for %Change from baseline values.

Produce similar tables for parameter Fractional excretion of sucralose.

Produce table for both the timepoints by page.

206243

Example PD\_T1
Protocol: 206243

Protocol: 206243 Page 1 of n
Population: Evaluable

Table 3.1
Summary of Intestinal Permeability/ Bacterial Translocation Associated Biomarkers

| Biomarkers(Unit) | Study Group | N | Visit | n | Mean | SD | SE | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| Claudin 3 | Healthy<br>Subjects | 200 | Day 1 | 200 | 91.6 | 11.32 | 0.80 | 90.0 | 68 | 140 |
| | TI<br>Subjects | 200 | Day 1 Day 3 Day 28 6 months | 200<br>190<br>195<br>186<br>195 | 91.6<br>92.4<br>92.1<br>92.6<br>92.1 | 11.32<br>9.83<br>10.80<br>10.87<br>10.80 | 0.80<br>0.71<br>0.77<br>0.80<br>0.77 | 90.0<br>90.0<br>89.0<br>89.0 | 68<br>70<br>72<br>69<br>72 | 140<br>122<br>120<br>125<br>120 |
| Citrulline | Healthy Subjects TI Subjects | 200 | Day 1 Day 1 Day 3 Day 28 6 months | 200<br>200<br>190<br>195<br>186<br>195 | 91.6<br>91.6<br>92.4<br>92.1<br>92.6<br>92.1 | 11.32<br>11.32<br>9.83<br>10.80<br>10.87<br>10.80 | 0.80<br>0.80<br>0.71<br>0.77<br>0.80<br>0.77 | 90.0<br>90.0<br>90.0<br>89.0<br>89.0 | 68<br>68<br>70<br>72<br>69<br>72 | 140<br>140<br>122<br>120<br>125<br>120 |

Note: Day 1 is considered as baseline for both the study groups.

#### Programming note:

Include all study visits for TI Subjects.

Produce same table for absolute, Change from baseline and % Change from baseline values for all biomarkers.


Example: EFF\_L1
Protocol: 206243

Population: Screened

Study Group: Healthy Subjects

Listing of Lactulose, Mannitol, L/M Ratio and Sucralose Data

| Site ID./ | Age(Y)/<br>Sex/ | 77 | Time | Date<br>/<br>Stud | Total<br>Volum<br>e of<br>Urine | uri<br>Lact | ne (Ur<br>Man | Sucr | Lact | action | Sucr | L/M | base<br>L/M | e from<br>line<br>Sucr | fr<br>base<br>L/M | Sucr |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subj | Race<br>Detail | Visi<br>t | poin<br>t | У<br>Day | (Unit | ulos<br>e | nit<br>ol | alos<br>e | ulos<br>e | Mann<br>itol | alos<br>e | rati<br>o | rati<br>o | alos<br>e | rati<br>o | alos<br>e |
| | | Day<br>1 | 0-5<br>hour<br>s<br>0-24<br>hour<br>s | 241 | , | ) | | | | 1001 | | | | | | |
| PPD | 57/ M/ Asian - Central /South Asian Heritag e | Day<br>8 | 0-5<br>hour<br>s<br>0-24<br>hour<br>s | | | | | | | | | | | | | |
| | υ | Day<br>15 | 0-5<br>hour<br>s<br>0-24<br>hour | | | | | | | | | | | | | |

206243

Example: PD\_L1

Population: Screened

Listing of Biomarker Data

| Study<br>Group | Site ID./<br>Subj. | Age(Y)/<br>Sex/<br>Race Detail | Biomarker<br>(Unit) | Visit | Date/<br>Study<br>Day | Character<br>result<br>[optional] | Numeric<br>Score | Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| | XXX/<br>XXX | 57/ M/<br>Asian -<br>Central/South<br>Asian Heritage | | Day 1 | | | | |
| | XXX/<br>XXX | | | | | | | |

206243

Example: TW\_L1
Protocol: 206243

Population: Screened


Listing of Time to Wound Recovery Data

| Study | Centre<br>ID./<br>Subj. | Age(Y)/<br>Sex/ | Visit | Screening<br>Date | Wound<br>recovery<br>Date | Time to wound recovery (in days) |
|---|---|---|---|---|---|---|
| Group | Subj. | Race Detail | VISIL | Date | Date | (III days) |
| | XXX/<br>XXX | 57/ M/<br>Asian -<br>Central/South<br>Asian Heritage | Day 1 | | | |
| | XXX/<br>XXX | | | | | |

Example: AG1


Population: Screened

### Listing of STM Administration

| Study<br>Group | Site ID./<br>Subj. | Age(YEAR<br>S)/<br>Sex/<br>Race<br>Detail | Visit | Start<br>date of<br>STM | Start<br>time of<br>STM |
|---|---|---|---|---|---|
| | | 57/ M/<br>Asian - | | | |
| | XXX/<br>XXX | Central/<br>South<br>Asian<br>Heritage | Day 1 | | |
| | XXX/<br>XXX | | | | |

206243

Example: SC1


Population: Screened

### Listing of Subject Characteristics

| Study<br>Group | Site ID./<br>Subj. id | Age(YEARS)/<br>Sex/<br>Race Detail | Subject characteristic | Result |
|---|---|---|---|---|
| | | | Subject ID for Non GSK Study | A-021 |
| | 3333 / | 57/ M/<br>Asian - | Recruited Within 24 Hr<br>Sustaining Injury | N |
| XXX/<br>XXX | Central/South<br>Asian<br>Heritage | Data and mine of David large | 21FEB2018T16:35 | |
| | | Date and Time of Enrollment | 20FEB2018T16:00 | |
| | | Date and Time of Injury | | |
| | XXX/ | | | |
| | XXX | | | |

206243

Example: SU3


Protocol: 206243
Population: Screened

Listing X
Listing of Substance Use

| Study<br>Group | Centre<br>id./<br>Subj. | Visit | Smoking<br>History | Last<br>smoked | Smokeless<br>Tobacco<br>History | Last used<br>Smokeless<br>Tobacco | Drink<br>Alcohol | Units<br>per<br>Week | Drink<br>Alcohol<br>Prior Study |
|---|---|---|---|---|---|---|---|---|---|
| Healthy<br>Subjects | PPD | Visit 1 | Never | | Never | | Yes | 20 | |
| | | Visit 1 | Current | | Current | | No | | |
| TI<br>Subjects | | Visit 1 | Former | 23JAN2016 | Never | | Yes | 15 | Yes,<br>21FEB2018<br>16:28 |


Example: EFF\_F1 Protocol: 206243

Population: Evaluable

Timepoint: 0-5 hours



Note: Above plot is based on healthy subjects.

Note: Reference line represents average over whole data for Healthy subjects which will be used as reference value for thermally injured Subjects.

Programming note: Include all the available Healthy Subjects in the plot. Produce this plot for endpoint L/M ratio and Sucralose. Produce similar graph for timepoint 0 – 24 hours.

Example: EFF\_F2
Protocol: 206243

Population: Evaluable






Note: Above plot is based on thermally injured subjects.

Note: The reference line (HSA) is based on average value of Healthy subjects.

Note: TI= thermally injured, HS=Healthy Subjects, S= thermally injured subject.

Programming note: Change HS to HSA in the legend in above graph. Include all the available TI subjects in the plot.

 $Produce\ similar\ plot\ for\ endpoint\ Sucralose.\ Also,\ produce\ graph\ for\ timepoint\ 0-24\ hours.$ 

The reference line for %CFB graph will be either 0 or average of %change in healthy subjects which will be decided based on the data.


Example: EFF\_F3
Protocol: 206243

Population: Evaluable

Timepoint: 0-5 hours

Figure x
Individual Plot of L/M Ratio and Sucralose Over Time for TI subjects



Note: D=Day, HS\_LM=Average value of L/M ratio based on healthy subjects, HS\_SL=Average value of Sucralose based on healthy subjects. Note: L/M Ratio and Sucralose raw values are based on thermal injured subjects.

Programming note: Produce similar graph for %CFB. Also, produce graph for timepoint 0-24 hours.

The reference line for %CFB graph will be either 0 or average of %change in healthy subjects which will be decided based on the data.

Example: PD\_F1
Protocol: 206243

Population: Evaluable


### Subject Profile plot for Intestinal Permeability/ Bacterial Translocation Biomarkers



206243

Note: Above plot is based on thermally injured subjects.

Note: The reference line (HSA: Healthy Subject's Average value) is based on average value of Healthy Subjects at day 1.

Note: HS= Healthy Subjects, S= thermally injured subjects.

Programming note: Include all the available thermally injured subjects in the plot.

Produce plot for all the biomarker groups.

Produce similar graph for %CFB.

The reference line for %CFB graph should be plot at 0.

Change HS to HSA in the legend in above graph.